CLINICAL TRIAL: NCT06032546
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-controlled Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of Budigalimab and/or ABBV-382 in People Living With HIV on Stable Antiretroviral Therapy Undergoing Analytical Treatment Interruption
Brief Title: A Study to Assess Change in Disease Activity, Adverse Events, and How the Drug Moves Through the Body in Adult Participants Living With Human Immunodeficiency Virus (HIV) Receiving Intravenous (IV) Infusion or Subcutaneous (SC) Injection of Budigalimab and/or ABBV-382
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-965; 2023-505900-53-00 (Other: EU CT)
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Human Immuno-deficiency Virus (HIV) Disease
Keywords: Human immuno-deficiency virus (HIV) Disease; Budigalimab; ABBV-382
MeSH Terms: conditions — Disease | interventions — budigalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Arm A: Placebo (Placebo Comparator): Participants will receive budigalimab placebo on Day 1, and Weeks 2, 4, and 6 in combination with ABBV-382 matching placebo on Day 1 and Weeks 4 and 8.
  Interventions: Drug: Placebo for Budigalimab; Drug: Placebo for ABBV-382
- Arm B: Budigalimab Dose A (Experimental): Participants will receive budigalimab Dose A on Day 1 and Weeks 2, 4, and 6 in combination with ABBV-382 matching placebo Day 1 and Weeks 4 and 8.
  Interventions: Drug: Budigalimab; Drug: Placebo for ABBV-382
- Arm C: ABBV-382 Dose A (Experimental): Participants will receive budigalimab placebo on Day 1 and Weeks 2, 4, and 6 in combination with ABBV-382 Dose A on Day 1 and Weeks 4 and 8.
  Interventions: Drug: Placebo for Budigalimab; Drug: ABBV-382
- Arm D: Budigalimab Dose A + ABBV-382 Dose B (Experimental): Participants will receive budigalimab Dose A on Day 1 and Weeks 2, 4, and 6 in combination with ABBV-382 Dose B on Day 1 and Weeks 4 and 8.
  Interventions: Drug: Budigalimab; Drug: ABBV-382
- Arm E: Budigalimab Dose A + ABBV-382 Dose A (Experimental): Participants will receive budigalimab Dose A on Day 1 and Weeks 2, 4, and 6 in combination with ABBV-382 Dose A on Day 1 and Weeks 4 and 8.
  Interventions: Drug: Budigalimab; Drug: ABBV-382
- Arm F: Budigalimab Dose B (Experimental): Participants will receive open-label budigalimab Dose B on Day 1 and Weeks 2, 4, and 6 (Note, no ABBV-382 or placebo will be administered).
  Interventions: Drug: Budigalimab

INTERVENTIONS:
Drug: Budigalimab — Intravenous (IV) Infusion
  Other Names: ABBV-181
  Arms: Arm B: Budigalimab Dose A; Arm D: Budigalimab Dose A + ABBV-382 Dose B; Arm E: Budigalimab Dose A + ABBV-382 Dose A
Drug: Placebo for Budigalimab — IV Infusion
  Arms: Arm A: Placebo; Arm C: ABBV-382 Dose A
Drug: ABBV-382 — IV Infusion
  Arms: Arm C: ABBV-382 Dose A; Arm D: Budigalimab Dose A + ABBV-382 Dose B; Arm E: Budigalimab Dose A + ABBV-382 Dose A
Drug: Placebo for ABBV-382 — IV Infusion
  Arms: Arm A: Placebo; Arm B: Budigalimab Dose A
Drug: Budigalimab — Subcutaneous (SC) Injection
  Other Names: ABBV-181
  Arms: Arm F: Budigalimab Dose B

SUMMARY:
Human immuno-deficiency virus (HIV) is the virus that causes Acquired Immuno-Deficiency Syndrome (AIDS). HIV disease is considered to be a chronic disease requiring lifelong therapy. The purpose of this study is to assess change in disease activity, adverse events, tolerability, and how the drug moves through the body.

Budigalimab and ABBV-382 are investigational drugs being developed for the treatment of HIV disease. In Part 1, participants are placed in 1 of 5 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 7 chance that participants will be assigned to placebo (A placebo is not a drug and it is not expected to have any chemical effects on your body and it is not designed to treat any disease or illness). In Part 2, eligible participants will be placed in an open-label arm to receive Budigalimab. Approximately 160 adult participants living with HIV disease on stable antiretroviral therapy (ART) willing to undergo Analytical Treatment Interruption (ATI) will be enrolled at approximately 90 sites worldwide.

In Part 1, participants will receive 4 doses of intravenous (IV) budigalimab or placebo combined with 3 doses of IV ABBV-382 or placebo for an 8 week dosing period. In Part 2, participants will receive 4 doses of open-label subcutaneous (SC) Budigalimab for a 6 week dosing period. Participants need to be stable on antiretroviral therapy to participate in the study. If participant qualifies to the study, on the day they receive the first injection, participants will be asked to stop antiretroviral medications (also referred to as analytical treatment interruption or ATI) for 112 weeks or until meeting specific criteria to restart antiretroviral medications. Participants will undergo a closely monitored ART interruption. Protocol-defined ART restart criteria includes participant's request. Participants will be followed for up to approximately 112 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. There will be an option for virtual or home health visits for some of the follow-up visits. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* A condition of general good health in the opinion of the investigator, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).
* Must be on antiretroviral therapy (ART) for at least 12 months prior to screening and on a stable ART regimen for at least 8 weeks prior to screening (current ART regimen cannot include an Non-nucleoside reverse transcriptase inhibitor [NNRTI] or long-acting ART).
* Negative human immuno-deficiency virus (HIV)-2 antibody (Ab)
* Cluster of differentiation 4 (CD4+) T cell count >= 500 cells/μL at screening and no known evidence of CD4+ T cell count < 500 cells/μL in the last 12 months prior to screening
* Participant must have plasma HIV-1 ribonucleic acid (RNA) below the lower limit of quantitation (LLOQ) at screening and for at least 12 months prior to screening

Exclusion Criteria:

* Prior exposure to long acting antiretrovirals within 24 weeks or within a period defined by 5 half-lives, whichever is longer, prior to randomization and prior to the first dose of study drug.
* History of CD4+ T cell nadir of <= 200 cells/μL during chronic HIV infection.
* History of medical disorders (other than HIV-1 infection) that, in the opinion of the investigator, might expose the participant to undue risk of harm, confound study outcomes or prevent the participant from completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Viral Control Without Antiretroviral Therapy (ART) Restart | Week 24
  Percentage of participants who achieve viral control (viral load < 1000 copies/mL) without ART restart at Week 24.
Number of Participants with Adverse Events (AEs) | Up to approximately Week 112
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Median Peak Viral Load (At Rebound) Prior to Re-Starting ART | Up to 112 weeks
  The median peak viral load (at rebound) before re-starting ART.
Median Time to First Rebound to >= 1000 Copies/mL During ART Interruption | Up to 112 weeks
  The median time to rebound to >= 1000 copies/mL during ART interruption.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (80):
- United States (43):
  - University of Alabama at Birmingham, 1917 Research Clinic /ID# 257549, Birmingham, Alabama
  - Franco Felizarta, Md /Id# 256927, Bakersfield, California
  - AHF Research Center /ID# 257025, Beverly Hills, California
  - Long Beach Education and Research Consultants /ID# 257552, Long Beach, California
  - AHF Healthcare Center- Hollywood /ID# 257026, Los Angeles, California
  - Los Angeles LGBT Center /ID# 258407, Los Angeles, California
  - Ruane Clinical Research Group /ID# 256932, Los Angeles, California
  - Palmtree Clinical Research Inc. /Id# 258409, Palm Springs, California
  - Optimus Medical /ID# 257182, San Francisco, California
  - Quest Clinical Research /ID# 256928, San Francisco, California
  - Washington Health Institute /ID# 259336, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center /ID# 257101, DeLand, Florida
  - AIDS Healthcare Foundation (AHF) - Healthcare Center - Northpoint /ID# 256934, Fort Lauderdale, Florida
  - Midway Immunology and Research Center /ID# 256930, Ft. Pierce, Florida
  - Advanced Pharma CR, LLC /ID# 259335, Miami, Florida
  - Orlando Immunology Center /ID# 256931, Orlando, Florida
  - Bliss Health /ID# 257827, Orlando, Florida
  - Baycare Medical Group - Tampa /ID# 256953, Tampa, Florida
  - The Pierone Research Institute /ID# 257022, Vero Beach, Florida
  - Triple O Research Institute /ID# 256929, West Palm Beach, Florida
  - Winship At Emory University Hospital Midtown /ID# 258410, Atlanta, Georgia
  - Metro Infectious Disease Consultants, P.L.L.C /ID# 256955, Decatur, Georgia
  - Howard Brown Health Center /ID# 257485, Chicago, Illinois
  - Claudia T. Martorell MD LLC dba The Research Institute /ID# 259155, Springfield, Massachusetts
  - KC CARE Health Center - Midtown South /ID# 257178, Kansas City, Missouri
  - Las Vegas Research Center /ID# 257619, Las Vegas, Nevada
  - Cooper University Health Care - Camden /ID# 258133, Camden, New Jersey
  - Saint Michael's Medical Center /ID# 258802, Newark, New Jersey
  - South Jersey Infectious Disease /ID# 257840, Somers Point, New Jersey
  - Unmhsc /Id# 257533, Albuquerque, New Mexico
  - Suny Upstate University Hospital Community Campus /ID# 257847, Syracuse, New York
  - Jacobi Medical Center /ID# 257849, The Bronx, New York
  - Montefiore Medical Center /ID# 257792, The Bronx, New York
  - East Carolina University - Brody School of Medicine /ID# 257544, Greenville, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 257542, Winston-Salem, North Carolina
  - Central Texas Clinical Research /ID# 256920, Austin, Texas
  - Prism Health North Texas - Oak Cliff Health Center /ID# 256933, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A /ID# 257592, Dallas, Texas
  - University of Texas Southwestern Medical Center /ID# 257551, Dallas, Texas
  - Texas Center for Infectious Disease Associates /ID# 257183, Fort Worth, Texas
  - The Crofoot Research Center, Inc /ID# 256921, Houston, Texas
  - DCOL Center for Clinical Research /ID# 257093, Longview, Texas
  - Wisconsin Medical Center /ID# 257498, Milwaukee, Wisconsin
- Belgium (4):
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 257433, Anderlecht, Brussels Capital
  - CHU Saint Pierre /ID# 257447, Brussels, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 257444, Brussels, Brussels Capital
  - UZ Gent /ID# 257446, Ghent, Oost-Vlaanderen
- Ricardo Diaz Scientific Solution /ID# 257335, São Paulo, São Paulo, Brazil
- Canada (6):
  - Spectrum Health Vancouver /ID# 260791, Vancouver, British Columbia
  - Ottawa Hospital Research Institute /ID# 256993, Ottawa, Ontario
  - Toronto General Hospital /ID# 256994, Toronto, Ontario
  - McGill University Health Centre - Glen Site /ID# 256992, Montreal, Quebec
  - CHU de Quebec-Université Laval hôpital CHUL /ID# 261611, Québec, Quebec
  - Regina General Hospital - Infectious Disease Clinic /ID# 260243, Regina, Saskatchewan
- France (2):
  - AP-HP - Hopital Saint-Antoine /ID# 258090, Paris
  - AP-HP - Hopital Tenon /ID# 258091, Paris
- Germany (3):
  - Infektiologikum /ID# 257112, Frankfurt am Main, Hesse
  - Universitaetsklinikum Bonn /ID# 257113, Bonn, North Rhine-Westphalia
  - zibp-Zentrum fuer Infektiologie /ID# 257110, Berlin
- Italy (4):
  - IRCCS Ospedale San Raffaele /ID# 259820, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 257410, Milan, Milano
  - Azienda Ospedaliera Universitaria Federico II /ID# 257412, Naples, Napoli
  - Azienda Ospedaliero-Universitaria di Modena /ID# 257411, Modena
- Japan (3):
  - NHO Nagoya Medical Center /ID# 261433, Nagoya, Aichi-ken
  - National Hospital Organization Osaka National Hospital /ID# 261520, Osaka, Osaka
  - IMSUT Hospital, The Institute of Medical Science, The University of Tokyo /ID# 265344, Tokyo
- Poland (2):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza /ID# 259184, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Punkt Zdrowia /ID# 257950, Gdansk, Pomeranian Voivodeship
- Puerto Rico (2):
  - Clinical Research Puerto Rico /ID# 256956, San Juan
  - HOPE Clinical Research /ID# 257487, San Juan
- South Africa (4):
  - Wits RHI Research Centre /ID# 257354, Johannesburg, Gauteng
  - Perinatal HIV Research Unit (PHRU) /ID# 257350, Johannesburg, Gauteng
  - Clinical HIV Research Unit (CHRU) /ID# 257358, Johannesburg, Gauteng
  - Ezintsha Research Centre /ID# 257391, Johannesburg, Gauteng
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol /ID# 257268, Badalona, Barcelona
  - Hospital Clinic de Barcelona /ID# 257269, Barcelona
  - Hospital Universitario Ramon y Cajal /ID# 257266, Madrid
  - Hospital Universitario La Paz /ID# 257170, Madrid
- United Kingdom (2):
  - Royal Free Hospital /ID# 257453, London, Greater London
  - Dup_Guys and St Thomas NHS Foundation Trust - Guy's Hospital /ID# 257761, London, Greater London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-965